CLINICAL TRIAL: NCT04184921
Title: A Multicenter, Prospective, Non-randomized, Open-label Study on the Efficacy and Safety of Osimertinib Combined With Aspirin as First-line Treatment for Patients With Locally Advanced or Metastatic EGFR-positive Non-small Cell Lung Cancer (NSCLC)
Brief Title: Combination of Osimertinib and Aspirin to Treat EGFR Mutation NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COAST 3
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer Non-small Cell Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aspirin; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osimertinib and aspirin (Experimental): Osimertinib and Aspirin starting at a dose of 80 mg and 100mg once a day, orally with meals. Aspirin treatment will be initiated one week before beginning TKI therapy, if possible, but TKI therapy will not be delayed for Aspirin loading. Drug: Osimertinib and Aspirin will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Interventions: Drug: Aspirin 100mg; Drug: Osimertinib 80 MG
- osimertinib (Active Comparator): Osimertinib starting at a dose of 80 mg once a day, orally with meals. Drug: Osimertinib will be administered once every day. If subject has complete response, partial response, stable disease, or unacceptable toxicity.
  Interventions: Drug: Osimertinib 80 MG

INTERVENTIONS:
Drug: Aspirin 100mg — Aspirin, also known as acetylsalicylic acid (ASA), is a very safe medication used to treat pain, fever, or inflammation.
  Arms: osimertinib and aspirin
Drug: Osimertinib 80 MG — Osimertinib, also known as azd9291, is a 3rd-generation EGFR-TKI used to treat NSCLC patients with resistance to 1st generation EGFR-TKI due to T790M mutation. It has been approved in clinical applications by the FDA in 2015.

SUMMARY:
The third generation epidermal growth factor receptor-tyrosine Kinase Inhibitor（EGFR-TKI） osimertinib has obvious curative effect for EGFR sensitive mutation and T790M mutation(PMID 27959700), but acquired drug resistance will occur. Previous studies show that apoptosis escape can lead to EGFR-TKI resistance.Osimertinib resistant cells show abnormal activation of PI3K/AKT/BIM activation(PMID 28765329). The classical drug aspirin can effectively decrease AKT phosphorylation and activate of BIM(PMID 28881293).So Investigators speculate that aspirin may decrease the PI3K/AKT/BIM signaling pathways, then promote osimertinib resistant cells apoptosis. The current study aims to evaluate the combination of aspirin and osimertinib in patients with EGFR/T790M mutations.

DETAILED DESCRIPTION:
Reversible small-molecule EGF receptor tyrosine kinase inhibitors (EGFR-TKI) have shown dramatic therapeutic efficacy in non-small cell lung cancer (NSCLC) patients with EGFR-activating mutations, and have been recommended as the standard first-line therapy in these patients. However, despite excellent initial clinical responses, nearly all patients eventually develop drug resistance after a median period of about 10 months(PMID 26497205). Osimertinib is a 3rd-generation EGFR-TKI used to treat NSCLC patients with resistance to 1st generation EGFR-TKI due to T790M mutation. But Osimertinib also face the problem of acquired drug-resistance(PMID 27959700). Thus, innovative treatment strategies are urgently needed to overcome therapeutic resistance to Osimertinib to improve the survival of patients with NSCLC.

Molecular mechanisms underlying acquired Osimertinib resistance are still not fully understood. Previous study showed that one principal mechanism accounting for majority of acquired resistance to Osimertinib in lung cancer is mediated by an exon 20 C797S mutation etc(PMID 29596911). More molecular mechanisms are still to be found. Apoptosis is a process of programmed cell death that occurs in multicellular organisms. Biochemical events lead to characteristic cell changes (morphology) and death. These changes include blebbing, cell shrinkage, nuclear fragmentation, chromatin condensation, chromosomal DNA fragmentation, and global mRNA decay. Apoptosis has been found to be related to drug resistance to 1st generation EGFR-TKI(PMID 29731879). The investigators previous found apoptosis is also related to Osimertinib resistance(PMID 28765329). Therefore, promoting apoptosis may be an effective way to improve the response to Osimertinib treatment.

Investigators' group has focused on lung cancer targeted therapy for several years. Previously, investigators have reported that metformin in combination with 1st generation EGFR-TKI could enhance the effect of TKI (PMID 24644001). Therefore, investigators further asked whether the drug combination approach could overcome osimertinib resistance. Aspirin is a widely used and well-tolerated drug for Kawasaki disease, pericarditis, and rheumatic and has arisen keen interest as a potential anticancer agent ever since the report of the clinical evidence that the cancer risk and mortality are reduced in Colon cancer. Aspirin exerts remarkable antitumor properties in tumor cells and mouse models. It strongly inhibited the growth of lung cancer cells, and its combination with TKI agents, including Sorafenib (PMID: 28857200), significantly suppressed RAS-mutant cancers growth and prolonged remission in a xenograft model. Interestingly, Aspirin exposure significantly promoted the apoptosis suggesting that aspirin may overcome Osimertinib resistance by promoting the apoptosis.

Here, investigators'group observed that in clinic, several patients who took osimertinib and aspirin together have shown excellent effect.Investigators therefore conduct this clinical trial to observe whether the combination of Aspirin and Osimertinib could enhance efficacy of Osimertinib in lung cancer patients with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

Locally advanced (stage IIIB) or metastatic (stage IV) EGFR-mutant NSCLC. Presence of EGFR-sensitive mutations suitable for treatment with Osimertinib. Intended to receive Osimertinib as first-line therapy, with an expected survival period of more than 3 months.

At least one measurable tumor lesion that meets the following criteria:

Not previously irradiated. Accurately measurable. Baseline longest diameter ≥10 mm (for non-lymph node lesions) or short axis ≥15 mm (for lymph node lesions).

Measurement can be performed via chest CT or PET-CT, provided the method allows reliable repeated measurements.

Exclusion Criteria:

Currently receiving other anticoagulant treatments. Patients planning to receive anticancer therapies other than Osimertinib. Presence of contraindications to the use of Osimertinib or Aspirin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival according to resist 1.1 | 5 years
  To evaluate the response to therapy and progression-free survival rate of the combination of Osimertinib and Aspirin in advanced lung cancer patients who has EGFR-mutation.

SECONDARY OUTCOMES:
overall survival（OS） | 5 years
  To evaluate the overall survival of the combination of Osimertinib and Aspirin in advanced lung cancer patients who has EGFR-mutation.
Objective Response Rate(ORR) according to resist 1.1 | 2 years
  To evaluate the response to therapy and Objective Response Rate of the combination of Osimertinib and Aspirin in patients who has EGFR-mutation.
Time to progression(TTP) according to resist 1.1 | 2 years
  To evaluate the response to therapy and Time to progression of the combination of Osimertinib and Aspirin in patients who has EGFR-mutation.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Result] Shi P, Oh YT, Deng L, Zhang G, Qian G, Zhang S, Ren H, Wu G, Legendre B Jr, Anderson E, Ramalingam SS, Owonikoko TK, Chen M, Sun SY. Overcoming Acquired Resistance to AZD9291, A Third-Generation EGFR Inhibitor, through Modulation of MEK/ERK-Dependent Bim and Mcl-1 Degradation. Clin Cancer Res. 2017 Nov 1;23(21):6567-6579. doi: 10.1158/1078-0432.CCR-17-1574. Epub 2017 Aug 1. PMID 28765329
- [Result] Ma J, Cai Z, Wei H, Liu X, Zhao Q, Zhang T. The anti-tumor effect of aspirin: What we know and what we expect. Biomed Pharmacother. 2017 Nov;95:656-661. doi: 10.1016/j.biopha.2017.08.085. Epub 2017 Sep 4. PMID 28881293
- [Result] Li L, Han R, Xiao H, Lin C, Wang Y, Liu H, Li K, Chen H, Sun F, Yang Z, Jiang J, He Y. Metformin sensitizes EGFR-TKI-resistant human lung cancer cells in vitro and in vivo through inhibition of IL-6 signaling and EMT reversal. Clin Cancer Res. 2014 May 15;20(10):2714-26. doi: 10.1158/1078-0432.CCR-13-2613. Epub 2014 Mar 18. PMID 24644001
- [Result] Li S, Dai W, Mo W, Li J, Feng J, Wu L, Liu T, Yu Q, Xu S, Wang W, Lu X, Zhang Q, Chen K, Xia Y, Lu J, Zhou Y, Fan X, Xu L, Guo C. By inhibiting PFKFB3, aspirin overcomes sorafenib resistance in hepatocellular carcinoma. Int J Cancer. 2017 Dec 15;141(12):2571-2584. doi: 10.1002/ijc.31022. Epub 2017 Sep 14. PMID 28857200